CLINICAL TRIAL: NCT02018029
Title: Predictives Factors of Cardiac Resynchronization Therapy: a Multimodal Analysis Using 2D Speckle Tracking Echocardiography Coupled With MIBG Myocardial Scintigraphy and Heart Failure Biomarkers
Acronym: PREFAC-CRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: General Electrics France (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-0173
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Heart Failure; Reduced Ejection Fraction
Keywords: Heart failure; Cardiac Resynchronisation Therapy; collagen peptides; MIBG scintigraphy
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

GROUPS / COHORTS (1):
- cardiac resynchronisation therapy
  Interventions: Other: cardiac resynchronisation therapy

INTERVENTIONS:
Other: cardiac resynchronisation therapy

SUMMARY:
Cardiac resynchronization therapy (CRT) is one of the lastest recommended treatments in patients with refractory symptomatic chronic heart failure with reduced ejection fraction (HFREF). Despite clear guidelines 20 to 40 % of implanted patients are not clinically ameliorated. They are called the "non responders". Patient selection seams to be one of the key to improve the efficiency of CRT. This protocol try to assess positive predictive factors to CRT by a multimodal approach.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) is a validated HFREF therapy. Unfortunately 20 to 40 % of implanted patients according to the guidelines do not have an improvement in their condition. The detection of "non responders" is imperfect. The selection of eligible patients to cardiac resynchronization is defined by symptomatic patients (NYHA class II to IV), a reduced Left Ventricle ejection fraction and by the duration of the left bundle branch block. No other parameter (clinical, electrical, echocardiographical) have been identified as positive predictive factor to cardiac resynchronization therapy.

The aim of the investigators study is to identify positive predictive parameters to CRT.

The investigators study included all patients eligible to CRT according to the guidelines of the European Society of Cardiology in four French centers (Clermont-Ferrand, Bordeaux, Nancy, Pasteur Toulouse).

1. At baseline a preimplantation evaluation is performed: clinical examination, laboratory assay (biological collection), echocardiography-2D Strain at rest and stress, myocardial perfusion scintigraphy and MIBG.
2. At 6 months, response to CRT is the primary endpoint. It is a composite primary endpoint, including modification of: Quality of Life Score (MINNESOTA scale) , NYHA functional status , 6-minute walk test and volume of the left ventricle. Three hundred patients are expected over a period of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 year's old
* Patient eligible to CRT according guidelines of ESC 2012:

QRS ≥ 120 ms and LVEF ≤ 35% and appearance typical block left arm and NYHA III and IV in sinus rhythm, QRS ≥ 150 ms and LVEF ≤ 35 % non- appearance block left leg NYHA III and IV in sinus rhythm, QRS ≥ 130 ms and LVEF ≤ 30% and appearance typical of LBBB NYHA II

* Life expectancy expected to exceed one year with a good functional status
* Optimal pharmacological treatment of heart failure

Exclusion Criteria:

* Pregnancy
* Contraindications to the CRT
* Fast atrial fibrillation
* Taking a treatment interfering with the binding of MIBG and can not be interrupted before the scan
* Contraindications to performing a scan [Hypersensitivity to the active substance (2-methoxy-isobutyl-isonitrile-(99mTc)and Iobenguane-(123l)) or any of the excipients, Pregnancy, Breastfeeding]
* Contraindication to achieve an uncontrolled stress test [Myocardial infarction in acute or very recent, unstable angina, prevent ventricular ejection (aortic stenosis, pulmonary stenosis, obstructive cardiomyopathy), severe hypertension, ventricular arrhythmia, and in all cases where it may be poorly tolerated : severe anemia , respiratory insufficiency, peripheral arterial disease, inability to walk or cycle ... ]
* No affiliation to the French social security system
* Refusal to participate
* Incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient eligible to cardiac resynchronisation therapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Composite primary endpoint | day of inclusion
  to evaluate response to CRT, modifications in NYHA class, 6-MWT, LV volumes and QOL scale.

SECONDARY OUTCOMES:
Mortality from any cause | at 6 months
Cardiovascular Mortality | at 6 months
Hospitalization for heart failure | at 6 months
Mortality from heart failure | at 6 months
Hospitalization for other cardiac causes | at 6 months
Hospitalization for all causes | at 6 months
Sudden Death recovered | at 6 months
Use of vasoactive amines | at 6 months
Cardiac Transplantation | at 6 months
Test of 6-minute walk | at 6 months
NYHA Class | at 6 months
Quality of life ( MINNESOTA ) | at 6 months
Change in systolic and / or diastolic left ventricular volume greater than or equal to 15% off between the two periods | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Romain ESCHALIER, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France